CLINICAL TRIAL: NCT04520360
Title: A Single-Center, Open-Label,Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of a New Oral Suspension and Tablet Formulation of Carisbamate (YKP509) in Healthy Adult Subjects
Brief Title: Bioavailability and Food Effect Study of 3 Types of Carisbamate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YKP509C005
Record Dates: First submitted 2020-08-05; First posted 2020-08-20 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: Carisbmate; Lennox-Gastaut syndrome (LGS); Healthy Volunteers
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, randomized, 5-period, 10-sequence study designed to assess each treatment in all subjects enrolled in the study. The five treatments tested using a single oral administration will be: (1) Oral Suspension Type 1, 300 mg Oral Tablet, Oral Suspension Type 2 all under fasted conditions and (2) Oral Suspension Type 2, 300 mg Oral Tablet under fed conditions. Each dose is followed by at least a seven-day washout period. The sequence and period arrangement will be constructed based on the Williams design to ensure the study is balanced with respect to first-order carry-over effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Types of Carisbamate (Experimental): 1. A single 300 mg oral dose of the Oral Suspension Type 1 under fasting conditions
  2. A single 300 mg oral dose of Oral Suspension Type 2 under fasting conditions
  3. A single 300 mg oral dose of Oral Suspension Type 2 under fed conditions
  4. A single oral dose of the 300 mg Oral Tablet under fasting conditions
  5. A single oral dose of the 300 mg Oral Tablet under fed conditions
  Interventions: Drug: Carisbamate

INTERVENTIONS:
Drug: Carisbamate — Carisbamate is currently under investigation as an adjuvant antiepileptic therapy in Lennox-Gastaut patients. Lennox-Gastaut syndrome (LGS) is a rare and highly debilitating form of childhood epilepsy that typically is diagnosed between 2 and 8 years of age, with peak onset at 3 to 5 years of age, and frequently persists into adulthood. Treatment options are limited and complicated by the multiple seizure types associated with LGS. Given the breadth of physical and cognitive disabilities associated with LGS, the development of antiseizure medications with appropriate oral dosing forms is needed to ensure administration feasibility and compliance in the target population.
  Other Names: YKP509

SUMMARY:
This study is designed to examine the relative bioavailability of three carisbamate formulations (Oral Suspension Type 1, Oral Suspension Type 2, and a 300 mg Oral Tablet) and to assess the effect of food on the oral bioavailability of the Oral Suspension Type 2 and the 300 mg Oral Tablet.

DETAILED DESCRIPTION:
This is a single center, open-label, randomized, 5-period, 10-sequence study designed to assess each treatment in 30 healthy subjects enrolled in the study. The five treatments tested using a single oral administration will be: (1) Oral Suspension Type 1, 300 mg Oral Tablet, Oral Suspension Type 2 all under fasted conditions and (2) Oral Suspension Type 2, 300 mg Oral Tablet under fed conditions. Each dose is followed by at least a seven-day washout period. The sequence and period arrangement will be constructed based on the Williams design to ensure the study is balanced with respect to first-order carry-over effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of 18 to 50 years of age (inclusive)
2. Able to read, understand, sign, and date a written informed consent form (ICF) before study participation at screening
3. Agree to use 2 highly effective methods of contraception, including at least one barrier method
4. Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening
5. Judged to be in good health based on medical history, physical examination, and routine laboratory measurements (i.e., without clinically relevant pathology)
6. Normal electrocardiogram (ECG) (12-lead), arterial blood pressure, and heart rate within the normal standard range used by the study center or considered not clinically significant by the Investigator and in agreement with the Sponsor
7. Able to understand and comply with protocol requirements and instructions and likely to complete the study as planned
8. A female study subject of childbearing potential must agree to use one of the accepted contraceptive method from Screening, during the study, and for at least 90 days after the last dose of the study medication. Hormonal contraceptives alone will not be considered an adequate method of contraception.
9. A female study subject must agree not to donate eggs (oocytes) during the study and for at least 90 days after the last dose of the study medication
10. Females of non-childbearing potential who have undergone a sterilization procedure at least 6 months prior to dosing with official documentation (e.g., hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy, hysterectomy, or bilateral oophorectomy) or become postmenopausal with amenorrhea for at least 1 year prior to dosing and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Principal Investigator's judgment
11. Subjects are able and willing to consume a high-fat meal within a 30 minute timeframe

Exclusion Criteria:

1. History of any illness or condition that, in the opinion of the Investigator, might confound the results of the study or pose additional risks in administering study drug to the subjects

1. Smokers (subjects who have smoked within 6 months prior to screening or those subjects with a positive result from the smoking screening assay)
2. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with pharmacokinetics of the study drug (except appendectomy and simple hernia repair).
3. Regular treatment with prescription medications. Subjects should have ended any prescription medications at least 14 days before the first dosing of the study drug. Potential subjects should only stop any prescribed medication at the direction of a physician or qualified medical professional.
4. Regular treatment with nonprescription medications. Subjects should have ended any nonprescription medications at least 14 days before the first dosing of the study drug. Potential subjects should consult with a physician or qualified medical professional before stopping any regular treatment with nonprescription medication.
5. Consumption of herbal medications, dietary supplements, and specific fruit products. Subjects should have stopped consumption of herbal medications or dietary supplements (e.g., St. John's Wort, ginkgo biloba, and garlic supplements), vitamins, and grapefruit or grapefruit juice, or Seville oranges at least 14 days before the first dosing of study drug.
6. History of drug or alcohol abuse or addiction within 2 years before the start of study drug dosing, or a positive test results for alcohol or drugs of abuse, such as amphetamine, barbiturate, benzodiazepine, cocaine, methadone, opiates, oxycodone, phencyclidine, propoxyphene, cannabinoid (THC), MDMA (Ecstasy), methaqualone, and tricyclic antidepressant (TCA).
7. Regular consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) before screening. Subjects may not consume any alcohol from 72 hours before the first dosing of study drug through the completion of the last PK sampling.
8. Consumption of an average of more than 5 servings per day of coffee, tea, chocolate, cola, or other caffeinated or methyl xanthine beverages before screening. Subjects may not consume any tea, coffee, chocolate, and other foods and beverages containing caffeine and other methyl xanthine derivatives from 48 hours prior to dosing until the collection of the last PK sample.
9. Participation in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 7 half-lives (whichever is longer) before screening.
10. Blood donation or a significant loss of blood within 60 days of the start of study drug dosing or donation of more than 1 unit of plasma within 7 days before screening.
11. Positive result at screening for any of the following infectious disease tests: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antigen and antibody (HIV-1/2 Ag/Ab)
12. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold])
13. History of any known relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
14. Women who are pregnant or breastfeeding
15. Subject who is judged not eligible for study participation by Investigator
16. Subject is at imminent risk of suicide (positive response to question 4 or 5 on the C-SSRS) or had a suicide attempt within 6 months prior to the Screening visit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 35 days
  To evaluate the safety and tolerability of each carisbamate formulation administered under either fed (Oral Suspension Type 2 and the 300 mg Oral Tablet) or fasted (all formulations) conditions. Evaluation of any abnormal laboratory safety results, ECGs or other incidence of treatment-emergent adverse events will be monitored. Subjects will also be assessed on the risk for suicidality via the C-SSRS (Columbia Suicide Severity Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Ry R Forseth, Ph.D., Study Chair — SK Life Science, Inc.
Locations (1):
- PRA Health Sciences- Salt Lake City, Salt Lake City, Utah, United States